CLINICAL TRIAL: NCT07065006
Title: Comparison of the Effects of Local Anesthetic Infiltration and Erector Spinae Plan (ESP) Block on Postoperative Recovery Quality and Pain in Lumbar Spinal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SINEM SARI, prof.dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025-150; 2025-150 (Other: Adnan Menderes University)
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Quality of Recovery and Pain Management
Keywords: wound local anesthetic infiltration; Erector Spinae Area (ESP) Block; quality of postoperative recovery; lumbar spinal surgeries
MeSH Terms: conditions — Agnosia; Bites and Stings

STUDY DESIGN:
Intervention Model Description: The study was designed as a double-blind, prospective randomized controlled trial.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esp (Other): After anesthesia and surgical intervention, bilateral ESP will be extended with ultrasound guidance from the midline 3 cm lateral at the T10 level. After the area is cleaned with povidone iodine before the block, the T10 transverse parts will be determined using a linear ultrasound probe. Local anesthetic will be applied to the erector spinae muscle with the needle used for peripheral block procedures and the transverse processor. Without administering local anesthesia, the location of the needle will be verified with the hydrodissection method with serum. After the location of the needle is verified, 20 ml of LA and a different mixture of serum will be changed and the same procedure will be repeated in the contralateral. 20 ml of the total 40 ml of LA will be bupivacaine 0.5%, which can be seen in 20 ml of serum.
  Interventions: Diagnostic Test: Qor-40 test (The recovery quality test); Other: Calculation of postoperative opioid consumption
- wound LAI (Other): For patients assigned to wound infiltration, 40 mL (20 ml of the total 40 ml of LA will be bupivacaine 0.5%, which can be seen in 20 ml of serum) will be infiltrated on both sides of the wound edges after closure.
  Interventions: Diagnostic Test: Qor-40 test (The recovery quality test); Other: Calculation of postoperative opioid consumption

INTERVENTIONS:
Diagnostic Test: Qor-40 test (The recovery quality test) — Scale of postoperative recovery quality at first 24th hour. Minimum score is 40=bad ,maximum score is 200=good
Other: Calculation of postoperative opioid consumption — Postoperative opioid consumptions on the pca (patient controlled analgesia) device of the patients will be recorded in Postoperative 30.min,1.,6.,12.,24. Opioid consumptions on the pca device of the patients will be recorded in 30.min,1.,6.,12.,24. hours.

SUMMARY:
Comparison of the Effects of Local Anesthetic Infiltration and Erector Spinae Plan (ESP) Block on Postoperative Recovery Quality and Pain in Lumbar Spinal Surgery

DETAILED DESCRIPTION:
The study was designed as a double-blind, prospective randomized controlled study. Blindness; healthcare professionals who will monitor the patient's pain in the postoperative period will not know whether ESP or wound local anesthetic infiltration block was applied. Randomization of the patients was planned to be done using computer support. It was planned to include 44 participants in the ESP block and wound local anesthetic infiltration groups. The current pain status of the patients in the ESP block and wound local anesthetic infiltration groups in the postoperative period will be evaluated with NRS (Numerical rating scale) at certain time intervals (30th min, 1st, 6th, 12th, 24th hour) during rest and movement. When the patients' NRS scores are 4 and above, intravenous analgesic will be administered additionally and the number of bolus doses of the patients with PCA in the first 24 hours will be recorded. The recovery quality of the patients who underwent both ESP block and RLB block at the postoperative 24th hour will be evaluated with the scoring system (QoR-40). Additionally, the patients' hemodynamic values will be recorded during these intervals.

ELIGIBILITY:
Inclusion Criteria:

* Elective lumbar surgery performed ASA I-III 18-75 years old

Exclusion Criteria:

1. Refusal at enrollment
2. Request for withdrawal from the study
3. Inability to give informed consent
4. Emergency surgery
5. Bleeding diathesis
6. Presence of contraindications to the LA agents used in this study
7. Use of chronic opioids
8. Psychiatric disorders
9. Presence of infection at the injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-07-10 (Estimated); Study Completion 2026-08-10 (Estimated)

PRIMARY OUTCOMES:
Qor-40 test (The recovery quality test) | 24th hour
  scale of postoperative recovery quality at first 24th hour. Minimum score is 40=bad ,maximum score is 200=good

SECONDARY OUTCOMES:
Postoperative opioid consumption | 30 minutes,1st hour,6th hour,12th hour and 24th hour
  Postoperative opioid consumptions on the pca (patient controlled analgesia) device of the patients will be recorded in Postoperative 30.min,1.,6.,12.,24. Opioid consumptions on the pca device of the patients will be recorded in 30.min,1.,6.,12.,24. hours.

IPD SHARING:
Plan to Share IPD: Undecided